CLINICAL TRIAL: NCT06116240
Title: A Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of TQB2450 Injection Combined With AL2846 Capsules in Patients With Advanced Solid Tumors
Brief Title: A Clinical Trial of TQB2450 Injection Combined With AL2846 Capsules in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-AL2846-I-01
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Pemetrexed; Injections; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Subjects with advanced hepatocellular carcinoma (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule
- Advanced gastric adenocarcinoma / gastroesophageal junction adenocarcinoma subjects (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule
- Advanced non-small cell lung cancer (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule
- Locally advanced or metastatic urothelial cancer (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule
- Advanced esophageal squamous cell carcinoma (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule
- Non-scaly and non-small cells lung cancer (Experimental): TQB2450 injection, 21 days as a treatment cycle. AL2846 capsule, 21 days as a treatment cycle. Pemetrexed disodium for injection, 21 days as a treatment cycle. Cisplatin injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection; Drug: AL2846 capsule; Drug: Pemetrexed disodium for injection; Drug: Cisplatin injection

INTERVENTIONS:
Drug: TQB2450 injection — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1).
Drug: AL2846 capsule — AL2846 is a multi-targeted tyrosine kinase receptor inhibitor
Drug: Pemetrexed disodium for injection — Pemetrexed disodium is a multi-target antifolate antineoplastic drug.
  Arms: Non-scaly and non-small cells lung cancer
Drug: Cisplatin injection — Cisplatin is a chemotherapy drug.
  Arms: Non-scaly and non-small cells lung cancer

SUMMARY:
This is a Phase Ib clinical trial to evaluate the safety and efficacy of TQB2450 injection combined with AL2846 capsules in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years old; Eastern Cooperative Oncology Group (ECOG) score: 0~1 point; Expected survival is more than 3 months;
* Subjects diagnosed by histopathological or cytology with hepatocellular carcinoma or gastric adenocarcinoma/adenocarcinoma of the gastroesophageal junction or non-small cell lung cancer or urothelial carcinoma or esophageal squamous cell carcinoma;
* Patients with hepatocellular carcinoma need to meet the following criteria at the same time:

  1. Previous treatment failure with at least one anti-angiogenic drug (such as sorafenib, lenvatinib, donafenib, bevacizumab, etc.) and one immune checkpoint inhibitor (such as PD-1, etc.);
  2. Subjects with Barcelona clinical liver cancer stage (BCLC stage) of stage C, or stage B subjects who are not suitable for local therapy or refractory to local therapy and are not suitable for radical treatment;
* Patients with advanced gastric adenocarcinoma/gastroesophageal junction adenocarcinoma who are not suitable for surgery and who have failed first-line standard chemotherapy (treatment of not less than 2 cycles) must meet any of the following criteria:

  1. disease progression occurs during first-line treatment, or disease progression occurs within 4 months after the last dose (including mono-therapy maintenance for first-line therapy) after the end of treatment;
  2. recurrence or metastasis during neoadjuvant or adjuvant therapy or within 6 months after the last dose is considered to be a failure of first-line systemic chemotherapy for advanced disease;
* Central nervous system (CNS) metastasis with no clinical symptoms or is accompanied by clinical symptoms, but the condition is controlled after treatment and the stability time is ≥ 4 weeks (subjects with central nervous system metastases need to be excluded from cohorts 4 and 6);
* Subjects with advanced non-small cell lung cancer must meet the following conditions:

  1. non-small cell lung cancer subjects who meet stage III.B/III.C/IV;
  2. previous failure of PD-1 inhibitors monotherapy or in combination with platinum-based chemotherapy;
* The previous treatment of patients with urothelial carcinoma meets any of the following:

  1. Those who can tolerate cisplatin chemotherapy have radiographically confirmed disease progression or recurrence during or after treatment;
  2. Those who cannot tolerate cisplatin chemotherapy, but can use carboplatin, etc., and radiographically confirmed disease progression or recurrence occurs during or after treatment;
  3. Not suitable for platinum-containing chemotherapy;
* Patients with advanced esophageal squamous cell carcinoma failure with previous immune checkpoint suppression agents such as PD-1/PD-L1;

Exclusion Criteria:

* Previously diagnosed with fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc. by histology or cytology;
* Pathological histology classification is squamous cell carcinoma (adenosquamous carcinoma including squamous cell carcinoma), carcinoid tumor, undifferentiated carcinoma or other gastric cancer/gastroesophageal junction adenocarcinoma that cannot be classified;
* Subjects with gastric adenocarcinoma/gastroesophageal junction adenocarcinoma known to be human epidermal growth factor receptor 2 (HER2)-positive (patients with unknown HER2 status must be confirmed at the local hospital) shall be excluded, but HER2-positive patients with disease progression after trastuzumab treatment can be enrolled;
* Previous treatment with anti-angiogenic drugs such as cabozantinib, apatinib, lenvatinib, sorafenib, sunitinib, bevacizumab (except subjects with advanced hepatocellular carcinoma)
* History of hepatic brain;
* According to imaging examination, the main trunk of the portal vein has cancer thrombus invasion, inferior vena cava or heart involvement;
* Hepatitis B combined with hepatitis C or hepatitis D infection;
* Patients who are preparing for or have received organ transplantation in the past;
* Other malignant tumors within 5 years (except for cured basal cell carcinoma of the skin, prostate carcinoma in situ and carcinoma in situ of the cervix, etc.);
* Those with a variety of factors that affect oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
* Patients with moderate to severe ascites with clinical symptoms requiring repeated drainage; Patients with uncontrolled pleural effusion and pericardial effusion;
* Patients with any bleeding or bleeding events ≥ CTCAE grade 3 within 4 weeks before the first dose; Patients with arteriovenous thrombotic events, such as cerebrovascular accident (including transient ischaemic attack), deep vein thrombosis, and pulmonary embolism, within 6 months prior to the first dose, are allowed to be treated with low molecular weight heparin, and antiplatelet agents are contraindicated throughout the study period;
* Those who have previously received radiotherapy, chemotherapy, surgery, etc., within less than 4 weeks before the first dose of study drug, less than 5 half-lives of oral targeted drugs or less than 14 days of oral fluorouracils;
* There are unhealed wounds, fractures, active ulcers of the stomach and duodenum, persistent positive fecal occult blood, ulcerative colitis, etc., or other conditions that may cause gastrointestinal bleeding and perforation as determined by the investigators;
* Liver cancer subjects have a history of gastrointestinal bleeding within 6 months before the first dose; Patients with portal hypertension have a high risk of bleeding considered by the investigators, or have a red sign confirmed by gastroscopy or gastroscopy.
* Other factors that the investigator determines that the subjects are not suitable to participate in this study;
* Subjects with Epidermal Growth Factor Receptor (EGFR) mutation and known anaplastic lymphoma kinase (ALK) translocation (for Advanced non-small cell lung cancer);
* Central squamous cell carcinoma with large hemoptysis risk (for Advanced non-small cell lung cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline up to 96 weeks
  Proportion of subjects achieving complete and partial response

SECONDARY OUTCOMES:
The incidence of Adverse events (AE) | Baseline up to 96 weeks
  The proportion of subjects with adverse events (AE), severe adverse events (SAE) and abnormal laboratory examination indicators
The severity of Adverse events (AE) | Baseline up to 96 weeks
  The severity of adverse events (AE), severe adverse events (SAE) and abnormal laboratory examination indicators assessed by Common Terminology Criteria For Adverse Events (CTCAE) 5.0.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Inner Mongolia Baotou Steel Hospital, Baotou, Neimenggu
  - Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Fifth Central Hospital, Tianjin, Tianjin Municipality